CLINICAL TRIAL: NCT01359579
Title: A Phase 1, Open-label, Pharmacokinetic, Safety, and Tolerability Study of a Single Oral Dose of Varespladib Methyl in Subjects With Normal Renal Function, and Subjects With Mild, Moderate, or Severe Renal Impairment
Brief Title: A Study of the Pharmacokinetics and Safety of Varespladib in Subjects With Normal or Impaired Renal Function
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AN-CVD2213
Record Dates: First submitted 2011-05-19; First posted 2011-05-25 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Renal Impairment
Keywords: renal impairment; phase 1; healthy volunteers
MeSH Terms: conditions — Renal Insufficiency | interventions — varespladib methyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subjects with mild renal impairment (Experimental)
  Interventions: Drug: varespladib methyl
- Subjects with moderate renal impairment (Experimental)
  Interventions: Drug: varespladib methyl
- Subjects with normal renal function (Experimental)
  Interventions: Drug: varespladib methyl
- Subjects with severe renal impairment (Experimental)
  Interventions: Drug: varespladib methyl

INTERVENTIONS:
Drug: varespladib methyl — Single oral 500 mg dose

SUMMARY:
The purpose of this study is to compare and evaluate the pharmacokinetic characteristics and the safety of varespladib methyl in mild or moderate renal impairment patients and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females 18 years or older with a BMI of 18-40 kg/m2 inclusive.
* Regarding renal function, subjects will be classified as either normal or as suffering from mild,moderate or severe renal impairment. Classification of renal impairment will be estimated by the MDRD and Cockcroft-Gault formulae

Exclusion Criteria:

* Any disease, condition and/or chronic medications which might compromise the hematologic, cardiovascular, pulmonary renal, gastrointestinal, hepatic, or central nervous system; or other conditions that might interfere with the distribution, metabolism or excretion of study drug, or would place the subject at increased risk
* Evidence of significant respiratory, gastrointestinal or hepatic disease at screening
* Positive screen for hepatitis B surface antigen, or HIV
* Positive test in drugs of abuse screens or alcohol on admission to the clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Measure of blood and urine levels of varespladib in subjects with renal impairment in comparison to subjects with normal renal function | PK samples will be collected predose and 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48, and 72 hours postdose

SECONDARY OUTCOMES:
Safety measures to include adverse events and changes in clinical laboratory results | From admistration of study drug through follow-up on Day 8

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Investigator Site 101, Orlando, Florida
  - Investigator Site 102, Minneapolis, Minnesota
  - Investigator Site 103, Knoxville, Tennessee